CLINICAL TRIAL: NCT07106008
Title: Clinical Application of a Novel Radiolabeled Translocator Protein (TSPO) Targeted Small Molecular Probe in Neuroinflammation Imaging of Glioma
Brief Title: Radiolabeled TSPO Targeted Molecular Probe in Glioma
Status: Not yet recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20250624-08-KS-01
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Glioma (Any Grade) in the Brain
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Evaluate the clinical application value of the novel radiolabeled TSPO-targeted molecular probe Gallium [68Ga]-DOTA-HK-011 in inflammation imaging of glioma.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary subjects, patients, or their legal representatives must sign the informed consent form.
* There are no restrictions on the gender of volunteers; age must be between 18 and 75 years, inclusive.
* Other imaging examination methods (e.g., CT, MRI) show the presence of intracranial lesions.
* Patients with brain glioma who are scheduled for surgery or biopsy that will provide final pathological results.
* Patients must have a kidney GFR > 50 mL/min, ERPF > 280 mL/min, platelet count (PLT) > 75,000/μL, white blood cell count (WBC) > 3,000/μL, and alanine aminotransferase (ALT) and asparta.

Exclusion Criteria:

* Individuals with a history of allergy to drugs with similar chemical or biological components to TSPO, a history of atopy, or currently suffering from allergic diseases.
* Individuals currently participating in other drug clinical studies, or who have previously participated in any drug (excluding vitamins and minerals) clinical studies.
* Individuals with other difficult-to-control clinical conditions, such as HIV infection, hepatitis C virus infection, active hepatitis B, other severe chronic infections, or serious mental, neurological, cardiovascular, respiratory, or other systemic diseases.
* Red blood cell count (RBC) < 4×10^12/L, white blood cell count (WBC) < 3×10^9/L, hemoglobin < 110 g/L, platelet count (PLT) < 75×10^9/L.
* Significant liver and kidney function abnormalities, glomerular filtration rate (GFR) < 50 ml/min.
* Tumor burden involving more than 50% of the affected organ, or significant spinal cord compression.
* Expected survival time less than six months, or having received chemotherapy within the past six months.
* Individuals with severe acute comorbidities or severe refractory mental disorders.
* Pregnant or breastfeeding women (pregnancy defined as a positive urine pregnancy test).
* Individuals whose physical condition is unsuitable for radioactive examination.
* Other circumstances deemed unsuitable for participation in the trial by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited through hospital electronic records and community health certers
Sampling Method: Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax of lesion uptake value | Time Frame: 60min after administration